CLINICAL TRIAL: NCT03555123
Title: A Randomized, Double-blind, Multicenter, Parallel, Placebo-controlled Study l to Evaluate the Efficacy and Safety of Short-term Administration of SIMDAX in Patients With Acutely Decompensated Heart Failure : Korea Bridging Study
Brief Title: Evaluate the Efficacy and Safety of Short-term Administration of SIMDAX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YY_YYBRS001
Record Dates: First submitted 2018-05-24; First posted 2018-06-13 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Acute Decompensated Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIMDAX (Experimental): Levosimendan2.5mg/mL
  Interventions: Drug: Simdax
- SIMDAX Placebo (Placebo Comparator): Water for injection
  Interventions: Drug: Simdax

INTERVENTIONS:
Drug: Simdax — Levosimendan2.5mg/ml

SUMMARY:
A randomized, double-blind, Multicenter, parallel, placebo-controlled study

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy, safety and tolerability of intravenous infusion of Levosimendan for 24hrs in patients with ADHF who will be hospitalized with ADHF and continue to have symptom of dyspnea at rest(NYHA Class III or IV) despite with treatment of SOCs(include intravenous diuretics, vasodilators and/or positive inotropic drugs but except amrinone and milrinone) within 48hrs

Efficacy is measured by Clinical composite classification(Improved, No change, Worse), bio-marker(change of BNP and ST-2), Patient's Global Assessment, NYHA functional Classification, hospitalization period and renal function tests(change of creatinine, BUN and NGAL) Safety is measured by recording the incidence of adverse events(AEs), vital signs, clinical blood safety tests(biochemistry, hematology) and concomitant medications

ELIGIBILITY:
Inclusion Criteria:

1. Written, signed and dated informed consent by the patient or the patient's legally authorized representative.
2. Male and female patients over 18 years of age.
3. Patients with chronic heart failure who were diagnosed with acute decompensated heart failure
4. Hospitalization for with a primary or secondary diagnosis at admission of worsening heart failure within the 48 hours prior to start of study drug infusion. Symptoms of worsening heart failure must have been treated with IV diuretics Patients who have been hospitalized more than 48 hours may be enrolled if they fail to improve clinically to treatments administered during the first 48 hours (1)(following initial improvement) their clinical status deteriorates either spontaneously or following the withdrawal of intravenous medications.

(2) Infusion rates for continuous IV diuretics, inotropes and vasodilators must have been unchanged for at least 2 hours prior to baseline.

5.Left ventricular ejection fraction less than or equal to 35% as assessed using echocardiography, radionuclide ventriculography or contrast angiography within the previous 12 months 6.Dyspnea at rest at both screening and baseline, as assessed by the patient.

Exclusion Criteria:

1. Severe obstruction of ventricular outflow tracts such as hemodynamically significant uncorrected primary valve disease and restrictive or hypertrophic cardiomyopathy.
2. Patients scheduled to receive angioplasty, cardiac surgery, a LV assist device or a heart transplant within 3months after randomization.
3. Patients who have undergone cardioversion during the 4 hours prior to baseline or are expected to undergo cardioversion in the 5 days after baseline.
4. Patients who have undergone a cardiac resynchronization procedure within the 30 days of screening or are expected to undergo such a procedure within 3 months.
5. Patients who have received an IV diuretics dose (including or change in dose of a continuous diuretic infusion) within 2 hours of the baseline assessments.
6. Patients who are intubated or otherwise not able to comply with the pre-study assessments.
7. Stroke or TIA within 3 months prior to randomization.
8. Systolic blood pressure 90 mmHg or less at screening or baseline.
9. Heart rate 120 bpm or greater, persistent for at least 5 minutes at screening or baseline.
10. Serum potassium less than 3.5mmol/l or greater than 5.4 mmol/l.
11. Angina pectoris during the 6 hours before baseline.
12. Administration of amrinone or milrinone within 24 hours before start of study drug infusion.
13. Hypersensitivity to levosimendan or any of the excipients: Povidone, Citric acid, Ethanol
14. A history of Torsades de Pointes.
15. Severe renal insufficiency (serum creatinine > 450mol/l (5.0 mg/dl)) or on dialysis.
16. Significant hepatic impairment or elevation of liver enzymes to 5 times the upper limit of normal.
17. Acute bleeding or severe anemia (hemoglobin < 10g/dl or blood transfusion during current admission) or acute decompensation due to an active infection
18. Patients with low hemoglobin between 9-10g/dl may be
19. Enrolled provided there is no evidence of bleeding, no intention to transfuse blood, no identified cause for anemia other than renal insufficiency and if the severity of anemia is longstanding (documented hemoglobin +/-1 g/dl of screening value > 30 days prior).
20. History of severe chronic obstructive pulmonary disease or unstable bronchial asthma as evidenced by e.g. CO2 retention or ongoing use of oral, intravenous or intramuscular steroids
21. Patients with pneumonia or pneumothorax
22. Patients with non-cardiac respiratory distress
23. A person with a BNP level of less than 100pg/mL on screening for an organ laboratory test.
24. Active infected patients who need to have symptoms of fever over 38.5℃ or get an intravenous administration of septicemia or antimicrobial agents.
25. Pregnant and lactating women
26. Patients who take Investigational Product including other clinical study within screening 4 weeks.
27. In case of unsuitable patients who are participated in this study because of other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the Clinical Composite Classification(CCC) | 5day
  Assessment of the Clinical Composite Classification(CCC) using the Patients Global Assessment(PGA) at 5day after start of IV levosiemendan or Placebo infusion with WHF through 5dyas: Improved, Unchanged, Worse

SECONDARY OUTCOMES:
BNP | baseline to 24hr, 48hr, 72hr, and 5day
  Change from baseline in plasma BNP levels at 24hr, 48hr, 72hr, and 5day
ST2 | baseline to 24hr, 48hr, 72hr, and 5day
  Change from baseline in plasma ST2 at 24hr, 48hr, 72hr, 5day
NYHA | baseline to 5day
  New York Heart Association(NYHA) functional classification at 5 days.
hospitalization | 31day
  Length of intensive care unit and /or Coronary care unit stay for the index ADHF hospitalization
cardio-renal biomarkers | baseline to 24hr, 48hr, 72hr, and 5day
  Change from baseline in cardio-renal biomarkers (Creatinine, BUN, NGAL) at 24hr, 48hr, 72hr and 5day
Patient's Global Assessment | 6hr
  Patient's Global Assessment (PGA, 7-likert scale) at 6 hr.
  : Check rate of patients who responded with Moderate or Marked improvement
Patients Assessment | 6hr
  Patients Assessment of dyspnea(7-likert scale) at 6hr
  : Check rate of patients who responded with Moderate or Marked improvement
re-hospitalization | 30days
  Time to re-hospitalization due to heart failure after discharge
death. | 30days
  Time to CV death.
mortality | 30days
  All cause mortality through 30days

CONTACTS AND LOCATIONS:
Overall Officials: Suck-min Kang, MD.PhD., Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No